CLINICAL TRIAL: NCT04672109
Title: The Effects of Different Montages of Transcranial Direct Current Stimulation on Muscle Strength in Healthy Adults
Brief Title: The Effects of Different Montages of tDCS on Muscle Strength in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MU2020
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anodal-tDCS (Experimental): Anodal transcranial direct current stimulation (tDCS) will be applied for 20 mins. Anode on the primary motor area (M1) of dominant hemisphere and Cathode on the supraorbital area of non-dominant hemisphere. Current intensity is fixed at 2 mA and current will flow continuously. The scope of intervention is to investigate effect of tDCS on muscle strength.
  Interventions: Device: Transcranial direct current stimulation
- Cathodal-tDCS (Experimental): Cathodal transcranial direct current stimulation (tDCS) will be applied for 20 mins. Cathode on the primary motor area (M1) of non-dominant hemisphere and Anode on the supraorbital area of dominant hemisphere. Current intensity is fixed at 2 mA and current will flow continuously. The scope of intervention is to investigate effect of tDCS on muscle strength.
  Interventions: Device: Transcranial direct current stimulation
- Dual-tDCS (Experimental): Dual transcranial direct current stimulation (tDCS) will be applied for 20 mins. Anode on the primary motor area (M1) of dominant hemisphere and Cathode on the primary motor area of non-dominant hemisphere. Current intensity is fixed at 2 mA and current will flow continuously. The scope of intervention is to investigate effect of tDCS on muscle strength.
  Interventions: Device: Transcranial direct current stimulation
- Sham-tDCS (Sham Comparator): Dual transcranial direct current stimulation (tDCS) will be applied over C3-C4 or the motor area (M1) for 20 mins. Anode on dominant hemisphere, Cathode on non-dominant hemisphere. The scope of intervention is to investigate effect of tDCS on muscle strength.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Dual/Cathodal/Anodal/Sham tDCS will be applied in 2 mA, 20 mins. All experiments will be performed in random order for each subject.

SUMMARY:
To investigate the effects of different montages of tDCS on muscle strength in healthy adults

DETAILED DESCRIPTION:
Electrode montage or placement of tDCS over primary motor cortex can be categorized into unilateral (anodal or cathodal electrode over primary motor area) and bilateral tDCS (both anodal and cathodal electrode over the cortex). Previous studies reported benefits of different tDCS montages on muscle performance in healthy participants. However, there is no guideline for tDCS montages. This study aims to investigate immediate effects of different tDCS montages on muscle strength in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults
2. Age range between 18 - 60 years old
3. Right-handed dominant identified by the Edinburg Handedness Inventory
4. No recent muscle injuries of both limbs for a past 6-months

Exclusion Criteria:

1. Consumed caffeine within 24 hours prior the experiment
2. History of neurological symptoms i.e. seizures, weakness, loss of sensation or unclear history of pass illness
3. Present of metal implantation, intracranial shunt, cochlear implantation or cardiac pacemakers
4. Present of opened wound or infectious wound around scalp

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline muscle strength after tDCS | Baseline (Pretest) and 40 minutes ( posttest)
  Muscle strength will be measured in Newton by using a hand-held dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Wanalee Klomjai, PhD, Study Director — MU
Locations (1):
- Faculty of Physical Therapy, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No